CLINICAL TRIAL: NCT07329660
Title: The Impact of Different Preload Strategies on Hemodynamics During Anesthesia Induction in TAVR Patients
Brief Title: Crystalloid vs Colloid for Hemodynamics During Anesthesia Induction in TAVR Patients
Acronym: CHAIN-T
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, associate professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJH-A-20250824
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Transcatheter Aortic Valve Replacement; Hemodynamic Stability; Anesthesia Induction
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colloid (Experimental): 5 ml/kg of hydroxyethyl starch 130/0.4 electrolyte injection.
  Interventions: Drug: Hydroxyethyl starch 130/0.4
- Crystalloid (Active Comparator): 5 ml/kg of sodium lactate Ringer's solution is administered before anesthesia induction.
  Interventions: Drug: Lactate Ringer's Solution

INTERVENTIONS:
Drug: Hydroxyethyl starch 130/0.4 — 5 ml/kg of hydroxyethyl starch 130/0.4 electrolyte injection is administered by infusion pump over 15 minutes before anesthesia induction.
  Arms: Colloid
Drug: Lactate Ringer's Solution — 5 ml/kg of sodium lactate Ringer's solution is administered before anesthesia induction.
  Arms: Crystalloid

SUMMARY:
The purpose of this study is to evaluate whether the administration of 5 ml/kg of colloid solution prior to anesthesia induction, compared with 5 ml/kg of lactated Ringer's solution, can reduce hemodynamic fluctuations during the induction period (defined as the first 15 minutes after induction) in patients undergoing Transcatheter Aortic Valve Replacement (TAVR).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patients scheduled to undergo elective TAVR under general anesthesia;

Exclusion Criteria:

* Allergy to hydroxyethyl starch, its components, and/or sodium lactate Ringer's solution, or a history of colloidal allergy;
* Severe cardiac dysfunction (ejection fraction[EF] < 35%);
* Severe renal dysfunction (creatinine > 132 μg/L and/or requiring renal replacement therapy);
* Morbid obesity (body mass index[BMI] > 37.5 kg/m² or > 32.5 kg/m² with metabolic diseases);
* Severe hepatic dysfunction ;
* Severe electrolyte disturbances ;
* Patients with preoperative intracranial hypertension requiring dehydration therapy;
* Expected postoperative hospital stay < 24 hours;
* Patients scheduled for multiple surgeries during this hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2026-01-04 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) of mean arterial pressure changes from baseline during the induction period. | induction period, at an average of 15 minutes
  The AUC below baseline mean arterial pressure (MAP) is calculated as:
  ∑ (((Si - Sbaseline)+(Si-1 - Sbaseline))/2 × ΔX)
  where Sbaseline is the baseline MAP, Si is the MAP at the i-th minute (i = 1…15), and ΔX is the time interval between two measurements.

SECONDARY OUTCOMES:
Incidence of post-induction hemodynamic instability, defined as arterial pressure (MAP)< 65 mmHg or a decrease of more than 20% from baseline within 15 minutes after induction. | 15 minutes after induction
Intraoperative use of vasoactive drugs. | Intraoperative period, at an average of 2 hours
Sequential Organ Failure Assessment(SOFA )score on the first postoperative day | The first postoperative day, at 24 hours after surgery
Length of hospital stay. | The duration of the patient's hospitalization after the initial surgery, at an average of 5 days.
Proportion of patients admitted to the intensive care unit (ICU) after surgery | During the postoperative period prior to discharge (at an average of 5 days)
In-hospital all-cause mortality | During the postoperative period prior to discharge (at an average of 5 days)
All-cause mortality within 30 days postoperatively | 30 days after surgery
Proportion of patients receiving renal replacement therapy during the 30-day postoperative observation period | 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Dong, Study Chair — Air Force Medical University